CLINICAL TRIAL: NCT01558583
Title: A Comparison of the Effect of a Conjoint Analysis Based Values Clarification Exercise, Rating and Ranking Exercise, and Balance Sheet for Colorectal Cancer Screening and Prostate Cancer Screening Decision Making
Brief Title: Online Study of Colorectal Cancer and Prostate Cancer Screening Decision Making
Acronym: CARR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCRF-CARR2-11-0861
Record Dates: First submitted 2012-02-07; First posted 2012-03-20 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2012-07

CONDITIONS: Colorectal Cancer; Colon Cancer; Prostate Cancer
Keywords: Colon; Prostate; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rating and Ranking Group (Other): A group of individuals from the United States and Australia who complete a rating and ranking task.
  Interventions: Other: Rating and Ranking Task
- Discrete Choice Group (Other): A group of individuals from the United States and Australia who complete a discrete choice experiment task.
  Interventions: Other: Discrete Choice Task
- Balance Sheet Group (Other): Individuals from the United States and Australia who will complete an implicit values clarification task
  Interventions: Other: Balance Sheet Task

INTERVENTIONS:
Other: Rating and Ranking Task — Individuals who are randomized to the rating and raking arm will be asked to complete an informational task in a rating and ranking format. The task will help individuals clarify their opinions and preferences regarding colon cancer and prostate cancer screening.
  Arms: Rating and Ranking Group
Other: Discrete Choice Task — Individuals who are randomized to the rating and raking arm will be asked to complete an informational task in a discrete choice format. The task will help individuals clarify their opinions and preferences regarding colon cancer and prostate cancer screening.
  Arms: Discrete Choice Group
Other: Balance Sheet Task — Individuals who are randomized to the rating and raking arm will be asked to complete an informational task in a balance sheet format. The task will help individuals clarify their opinions and preferences regarding colon cancer and prostate cancer screening.
  Arms: Balance Sheet Group

SUMMARY:
Participants will be recruited from the United States and Australia to take an online survey about colon cancer screening or prostate cancer screening. Individuals selected for both the prostate cancer survey and the colon cancer study will be randomized to take one of three survey types - balance sheet, rating and ranking or conjoint analysis. These surveys will help participants clarify their values and opinions about screening options for colon cancer or prostate cancer. Participants' responses to the online survey are measured at one point in time - the time at which the participant takes the survey.

DETAILED DESCRIPTION:
This study will compare effect of a conjoint analysis based values clarification exercise, ranking and rating, and a balance sheet on screening test preferences for colorectal cancer screening and prostate cancer screening using online surveys. Recruitment will be conducted through Survey Sampling International (SSI), an online survey research firm. Participants will be randomized to one of three arms to take online surveys. Patients will complete either a conjoint analysis task, in which they will be asked to make a series of choices between hypothetical screening testing strategies with different attributes; a rating and ranking task for these same attributes; or they will make a choice after viewing a balance sheet of attributes.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer

  * men and women, ages 50-75, who can speak and read English.
* Prostate cancer screening

  * men, ages 50-75, who can speak and read English.

Exclusion Criteria:

* Colorectal Cancer

  * individuals with a previous personal or family history of colon cancer, personal history of polyps, or inflammatory bowel disease will be excluded.
* Prostate cancer

  * individuals with a previous personal or family history of prostate cancer will be excluded

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1831 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Participant-reported most important attribute from survey | 1 day
  The single most important colon cancer or prostate cancer screening attribute indicated by the participant surveys. Each participant will be randomly assigned to take one of three survey versions: either (1) a conjoint analysis task wherein they will be asked to make a series of choices between hypothetical screening testing strategies with different attributes; (2) a rating and ranking task for these same attributes; or (3) they will make a choice after viewing a balance sheet of attributes.

SECONDARY OUTCOMES:
Participant-reported intent to undergo screening from survey | 1 day
  the number of participants who state they plan to be screened for condition
Unlabeled screening test options | 1 day
  choice on a single question among unlabeled screening test options

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pignone, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Cecil G. Sheps Center for Health Services Research, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Brenner A, Howard K, Lewis C, Sheridan S, Crutchfield T, Hawley S, Reuland D, Kistler C, Pignone M. Comparing 3 values clarification methods for colorectal cancer screening decision-making: a randomized trial in the US and Australia. J Gen Intern Med. 2014 Mar;29(3):507-13. doi: 10.1007/s11606-013-2701-0. Epub 2013 Nov 23. PMID 24272830
- [Derived] Howard K, Brenner AT, Lewis C, Sheridan S, Crutchfield T, Hawley S, Nielsen ME, Pignone MP. A comparison of US and Australian men's values and preferences for PSA screening. BMC Health Serv Res. 2013 Oct 5;13:388. doi: 10.1186/1472-6963-13-388. PMID 24093428
- [Derived] Pignone MP, Howard K, Brenner AT, Crutchfield TM, Hawley ST, Lewis CL, Sheridan SL. Comparing 3 techniques for eliciting patient values for decision making about prostate-specific antigen screening: a randomized controlled trial. JAMA Intern Med. 2013 Mar 11;173(5):362-8. doi: 10.1001/jamainternmed.2013.2651. PMID 23400279